CLINICAL TRIAL: NCT01013766
Title: A Randomized, Open-Label Study to Evaluate the Safety,Tolerability, Pharmacokinetics, and Pharmacodynamics ofGSK1362885 in Subjects With Type 2 Diabetes Mellitus
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of GSK1362885 in Type 2 Diabetics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 111823
Record Dates: First submitted 2009-10-29; First posted 2009-11-16 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: GSK1362885; Pharmacodynamics; Safety; Pharmacokinetics; T2DM; Tolerability
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- AM/PM/BID (Other): Subjects will receive a dose of 100mg in the AM on Day 1, followed by a dose of 100mg in the PM on Day 4, and a dose of 50mg BID on Day 6.
  Interventions: Drug: GSK1362885
- PM/AM/BID (Other): Subjects will receive a dose of 100mg in the PM on Day 1, followed by a dose of 100mg in the AM on Day 4, followed by 50mg BID on Day 6.
  Interventions: Drug: GSK1362885

INTERVENTIONS:
Drug: GSK1362885 — 100mg in the AM, 100mg in the PM, 50mg BID
  Arms: AM/PM/BID
Drug: GSK1362885 — 100mg in the PM, 100mg in the AM, 50mg BID
  Arms: PM/AM/BID

SUMMARY:
This study is the second administration of GSK1362885 in humans. GSK1362885 is a novel, potent inhibitor of human glycogen phosphorylase (GP) under development for the treatment of type 2 diabetes mellitus (T2DM). This study will investigate the compound's safety, tolerability, pharmacokinetics, and pharmacodynamics in subjects with Type 2 Diabetes Mellitus.

DETAILED DESCRIPTION:
This is the first administration of single doses of GSK1362885 to the target population with T2DM. Based on the mechanism of action which involves reducing hepatic glucose output, it is possible that day time (AM) or night time (PM) dosing of GSK1362885 could produce different plasma glucose lowering effects, acting either on prandial or post-absorptive elevations of HGO. This study is designed to compare glucose profiles following AM and PM doses to determine if there is any advantage to either one. This study will compare glucose profiles following a single dose of GSK1362885 in the morning before breakfast (AM) to a single dose administered at night (PM). These two dosing periods will be randomized and each subject will receive both dosing regimens. A third dosing period (BID) is not randomized, but is included to explore the effects of GSK1362885 on glucose profiles when administered twice daily in a 24 hour timeframe.

ELIGIBILITY:
Inclusion Criteria:

A subject will be eligible for inclusion in this study only if all of the following criteria apply:

* A diagnosis of T2DM as determined by a responsible physician based on a medical evaluation including medical history, physical examination, and laboratory tests. Subjects may be entered if they have stable hypertension or hyperlipidemia on therapy. Subjects with other conditions except as noted in Exclusion Criteria may be included only if the Investigator and the GSK medical Monitor agree that the condition is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Male or female between 18 and 65 years of age, inclusive, at the time of signing the informed consent.
* A female subject is eligible to participate if she is of non-childbearing potential, defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal/premature ovarian failure defined as 12 months of spontaneous amenorrhea. FSH and estradiol levels will be checked at Screening for postmenopausal women. Simultaneous follicle stimulating hormone (FSH) greater than 40 MlU/ml and estradiol less than 40 pg/ml (<140 pmol/L) is confirmatory.
* BMI within the range 22 to 38 kg/m2 (inclusive).
* T2DM diagnosed at least 3 months prior to Screening with:
* Fasting plasma glucose (FPG) level less than or equal to 250mg/dL at the Screening visit,
* FPG level less than or equal to 270 mg/dL on Day -2
* For subjects taking no antidiabetic medications: HbA1c between 6.5 and 11 percent, inclusive, at Screening visit
* For subjects taking one or two antidiabetic medications: HbA1c between 5.8 and 10 percent, inclusive, at Screening visit
* Subjects must be treating their T2DM using one of the following regimens:
* Diet and exercise therapy
* Metformin as monotherapy
* Sulfonylurea as monotherapy
* Metformin and sulfonylurea in combination, if one or both component(s) is being administered at a dose that is less than the maximum dose
* DPP-IV inhibitors, either as monotherapy, or in combination with other agent(s) on this list, if one or both component(s) is being administered at a dose that is less than the maximum dose
* Exenatide, either as monotherapy or in combination with other agent(s) on this list, if one or both component(s) is being administered at a dose that is less than the maximum dose
* All doses of anti-diabetic medication must have been stable for at least 2 months prior to Screening, and the subject must be willing to wash out from their antidiabetic medications from Day -10 through Day 7.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

A subject will not be eligible for inclusion in this study if any of the following criteria apply:

* Has any of the following laboratory abnormalities:
* Positive pre-study Hepatitis B surface antigen or positive Hepatitis C result within 3 months of screening.
* Positive test for HIV antibody
* History of uncorrected thyroid dysfunction or an abnormal thyroid function test assessed by TSH at Screening. (NOTE: subjects with hypothyroidism on a stable dose of thyroid replacement therapy for at least 3 months prior to Screening and who have a screening thyroid stimulating hormone (TSH) within the normal range may participate.)
* A positive pre-study drug/urine screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines.
* A pre-study urine cotinine screen indicating use of tobacco/ nicotine containing products.
* Subjects with values outside the specified ranges for the following Key Clinical Laboratory Tests must be excluded from the study. Laboratory tests may be repeated once at the discretion of the investigator.
* Liver function tests: ALT, Direct Bilirubin, or Albumin more than 10 percent outside the normal reference range (less than 0.9 x LLN or greater than 1.1 x ULN)
* Electrolytes: Sodium more than 5mEq/L outside the normal reference range, Potassium or Calcium more than 10 percent outside the normal reference range (less than 0.9x LLN or greater than 1.1 x ULN)
* Fasting Total Cholesterol greater than 240mg/dL, or Triglycerides greater than 450mg/dL
* Muscle: CPK greater than 1.5 x ULN
* Hematology: Hemoglobin, WBC, Neutrophils, or Platelets more than 10 percent outside the normal reference range (less than 0.9 x LLN or greater than 1.1 x ULN)
* Significant renal disease as manifested by one or more of the following:
* Creatinine clearance less than 60 mL/min.
* Urine protein/creatinine (mg/mg) ratio greater than 2.5; or urine albumin concentration greater than 300 ug/mg of creatinine.
* Known loss of a kidney either by surgical ablation, injury, or disease
* Other Clinical Laboratory Tests, not listed as a Key Clinical Laboratory Tests in Exclusion Criterion #4, should also be considered by the Investigator in the overall evaluation of a subject's suitability for enrollment in the study.
* Significant ECG abnormalities as defined per protocol
* Resting systolic blood pressure less than 80 mmHg or greater than 150 mmHg or diastolic blood pressure less than 60 mmHg or greater than 95 mmHg at screening. Blood pressure assessments may be repeated once if needed, allowing adequate time for subject to rest.
* Previous use of insulin as a treatment within 3 months of Screening, or for greater than 2 weeks when used for acute illness in the last 12 months prior to Screening, or if used for more than 1 year when associated with GDM.
* Has a history of any of the following conditions:
* Clinically significant symptoms of gastroparesis.
* Cholelithiasis or obstructive or inflammatory gallbladder disease within 3 months prior to Screening.
* Gastrointestinal disease that could affect fat or bile acid absorption, including inflammatory bowel disease, chronic diarrhea, Crohn's or malabsorption syndromes within the past year.
* Gastrointestinal surgery surgery within the past 6 months for laparotomy or past 3 months for laparoscopy including cholecystectomy
* Chronic or acute pancreatitis within the past year.
* History of regular alcohol consumption averaging greater than 7 drinks/week for women or greater than 14 drinks/week for men. 1 drink is equivalent to (12 g alcohol) = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of 80 proof distilled spirits) within 6 months of screening.
* Smoked or used tobacco or nicotine-containing products within the previous 6 months.
* Has participated in a clinical trial and has received a drug or a new chemical entity within 30 days or 5 half-lives, or twice the duration of the biological effect of any drug (whichever is longer) prior to the first dose of current study medication.
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Is taking prohibited medications. See Section 9 for a detailed list of prohibited medications. Note also:
* The use of anti-diabetic agents other than those listed in Inclusion #6 is reason for exclusion and subjects will not be allowed to wash off of unapproved anti-diabetic medications in order to qualify for participation in this study.
* Subjects must wash out from the following medications during the 10-day period prior to first dose, and must remain off these medications through discharge on Day 7: all antidiabetic medications specified in Inclusion #6, all statin agents, fat absorption blocking agents, and bile acid sequestrants. Fibrates must be washed out for a 14-day period prior to first dose.
* Vitamins, herbal and dietary supplements (including St John's Wort) are prohibited within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study medication and through discharge on Day 7.
* Unwilling to abstain from
* Caffeine-or xanthine-containing products for 24 hours prior to dosing until Day 7
* Use of illicit drugs or nicotine-containing products
* Alcohol for 24 hours prior to dosing until Day 7
* Consumption of red wine, Seville oranges, grapefruit or grapefruit juice from 7 days prior to the first dose of study medication until collection of the final pharmacokinetic blood samples
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the physician responsible, contraindicates their participation. This includes sensitivity to heparin, if heparin will be used to maintain catheter patency.
* Where participation in the study would result in donation of blood in excess of 500 mL within a 56 day period.
* Subject is either an immediate family member of a participating investigator, study coordinator, employee of an investigator; or is a member of the staff conducting the study.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Individual or family history of glycogen storage disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2009-08-13 (Actual); Primary Completion 2009-11-20 (Actual); Study Completion 2009-11-20 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability assessments including adverse events and clinical laboratory tests | 7 Days
Pharmacodynamics following oral administration (glucose, insulin, c-peptide) | 24 hours
Pharmacokinetic parameters: AUC, Cmax, Tmax, t1/2, tlag, Cl/F, and V/F | 24 hours

SECONDARY OUTCOMES:
Pharmacodynamics following BID administration (glucose, insulin, c-peptide) | 24 hours
Relationship between pharmacokinetic and pharmacodynamic parameters | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- United States (2):
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Saint Paul, Minnesota

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 111823 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/111823?search=study&search_terms=111823#rs
- Available data/document: Study Protocol: 111823 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 111823 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 111823 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 111823 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 111823 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 111823 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 111823 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register